CLINICAL TRIAL: NCT01802229
Title: Prevention of Umbilical Port-site Hernia After Laparoscopic Cholecystectomy Using a Prosthetic Mesh Versus Simple Suture
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital General Universitario Elche (Other)
Responsible Party: Principal Investigator, Jaime Ruiz-Tovar, MD, PhD, Professor, Hospital General Universitario Elche
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2013-002
Record Dates: First submitted 2013-02-27; First posted 2013-03-01 (Estimated); Last update posted 2013-03-01 (Estimated); Status verified 2013-02

CONDITIONS: Port-site Hernia

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Suture (Active Comparator): Umbilical port-site closure with simple suture of the fascia.
  Interventions: Procedure: Fascial suture
- Prophylactic mesh (Experimental): Umbilical port-site closure with mesh placement
  Interventions: Procedure: Prophylactic mesh placement

INTERVENTIONS:
Procedure: Prophylactic mesh placement — Placement of a Omega 3 mesh, fixed to the border of the fascia
  Arms: Prophylactic mesh
Procedure: Fascial suture — The port-site hole is closed with simple suture of the fascia
  Arms: Suture

SUMMARY:
The incidence of port-site hernia in patients with risk factors (obesity, elderly, diabetes and lung disorders) can be reduced by the use of a prophylactic mesh in the closure of umbilical port site.

ELIGIBILITY:
Inclusion Criteria:

* Age > 65 years
* BMI > 30 Kg/m2
* Diabetes mellitus
* Lung disease
* Elective laparoscopic cholecystectomy

Exclusion Criteria:

* Umbilical hernia
* Previous laparotomy
* Conversion to open procedure
* Loss during the follow up

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2011-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Incidence of port-site hernia | 12 months
  Comparison of incidence of port-site hernia between patiensts with and without prophylactic mesh placement

SECONDARY OUTCOMES:
Postoperative pain | 12 months
  Evaluation of different pain perception in patients with and without prophylactic mesh placement, determined in the postoperative course and at 1, 6 and 12 months after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital general Universitario de Elche, Elche, Alicante, Spain